CLINICAL TRIAL: NCT01872416
Title: A Clinical Study of Liposomal Doxorubicin Combined With Ifosfamide Second-line Treatment in Small Cell Lung Cancer: Single Center, Single-arm Study
Brief Title: A Clinical Study of Liposomal Doxorubicin Combined With Ifosfamide Second-line Treatment in Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, The First Affiliated Hospital of Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAHG20120926A; FAHGuangzhou012 (Registry Identifier: FAHGuangzhou012)
Record Dates: First submitted 2013-05-17; First posted 2013-06-07 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Small Cell Lung Cancer
Keywords: Refractory and relapsed small cell lung cancer; Liposomal Doxorubicin; ifosfamide
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Refractory and relapsed SCLC (Experimental): Liposomal Doxorubicin Combined With ifosfamide Second-line Treatment in Small Cell Lung Cancer
  Interventions: Device: Liposomal Doxorubicin Combined With ifosfamide

INTERVENTIONS:
Device: Liposomal Doxorubicin Combined With ifosfamide — Liposomal Doxorubicin Combined With ifosfamide Second-line Treatment in Small Cell Lung Cancer

SUMMARY:
At present, there is no standard second-line treatment of refractory and relapsed SCLC, topotecan, gemcitabine, paclitaxel, irinotecan and drugs such as cyclophosphamide second-line treatment of small cell lung cancer currently being explored, Anthracycline antibiotics is a cell cycle non-specific anticancer drugs could inhibit the synthesis of DNA, DNA and dependent RNA, its wide antitumor spectrum, widely used in malignant hematologic diseases and lung cancer and other solid tumors. Jacot W, et al evaluated epirubicin combined with ifosfamide (EI) for treatment of refractory and recurrent SCLC in 70 cases, the objective response rate (ORR) reached 21.4%, including 1 cases of complete remission, 10% other patients obtained stable disease (SD), all the patients had a median survival of 3.9 months, most (71%) patients with neutropenia, platelet count and anemia are also common, showed that EI treatment of refractory and relapsed SCLC is effectively controlled, toxicity.

In view of epirubicin combined with ifosfamide (EI) scheme is effective and safety in the treatment of refractory and relapsed SCLC, the investigators will use liposomal doxorubicin plus ifosfamide second-line treatment of refractory and relapsed small cell lung cancer, may obtain better tumor remission rate, improve the prognosis of the patients.

DETAILED DESCRIPTION:
the investigators will evaluate the overall response rate (complete and partial responses) in first-line treatment failure or relapse after first-line therapy SCLC treated with Pegylated liposomal doxorubicin and ifosfamide We will evaluate the progression-free survival (PFS) and overall survival (OS) i in receiving first-line treatment failure or relapse after first-line therapy SCLC treated with Pegylated liposomal doxorubicin and ifosfamide

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients >=18 years of age
2. the histological diagnosis of small cell lung cancer;
3. Patients who had first-line treatment failure or relapse after first-line therapy;
4. enough tumor tissue specimens for molecular marker analysis;
5. Measurable disease by RECIST criteria
6. ECOG performance status of <=2.
7. Life expectancy of at least 3 months.
8. Laboratory values as follows:: ANC ≥ 1.5 × 109/L; platelet count ≥ 100 × 109/L; HB ≥ 90g/L; serum bilirubin ≤ 1.5 upper limit of normal (N); ALT/AST≤ 2N (in patients with liver metastases :ALT/AST≤ 5N) creatinine≤1.25 N;and clearance rate of creatinine ≥ 60mLl/min; proteinuria < 2+, or were detected in 24 hour urine protein, protein content is ≤1g
9. Patient must be accessible for treatment and follow-up
10. All patients must be able to understand the nature of the study and give written informed consent prior to study entry

Exclusion Criteria:

1. mixed small cell lung cancer;
2. patients had a previous diagnosis of malignant tumor;
3. HIV infection;
4. A history of cardiac disease as defined by malignant hypertension, unstable angina, congestive heart failure of > grade 2 per New York Heart Association (NYHA) criteria, myocardial infarction within the previous 6 months, or symptomatic cardiac arrhythmias.
5. patients had the motor or sensory neurons lesions/symptoms of NCI - CTC AE > 1;
6. patients had serious active infections;
7. patients were allergic to ifosfamide or liposomal doxorubicin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
objective response rate | From date of randomization until the date of progression, assessed up to 5 months
  participants will be followed for the duration of hospital stay, an expected average of 5 months

SECONDARY OUTCOMES:
progression free survival(PFS） | From date of randomization until the date of progression, assessed up to 5 months

OTHER OUTCOMES:
overall survival | From date of randomization until the date of death from any cause, assessed up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: jianxing He, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- he First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China